CLINICAL TRIAL: NCT02688192
Title: Teens Living With Cancer Fitness Improvement Training (TLCFIT): A Novel Mobile Health Fitness Program for Adolescent and Young Adult (AYA) Childhood Cancer Survivors
Brief Title: Mobile Health Fitness Program for Adolescent and Young Adult Childhood Cancer Survivors
Acronym: TLCFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Katie Devine, PhD, MPH, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2013003658; NCI-2015-01841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 131323 (Other: Rutgers Cancer Institute of New Jersey); K07CA174728 (NIH); P30CA072720 (NIH)
Record Dates: First submitted 2015-11-30; First posted 2016-02-23 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Survivorship; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Intervention) (Active Comparator): Assessment including
  1. Wear an electronic accelerometer
  2. Quality of life assessment
  3. Physical fitness evaluation
  4. Participate in a fitness program which includes:
     * 8 group meetings of 90 minutes weekly
     * Behavioral internet based intervention engage in private social support messaging within the app and Facebook private groups and mobile app
  Interventions: Behavioral: Exercise Intervention; Behavioral: Internet-Based Intervention; Device: Monitoring Device; Other: Quality-of-Life Assessment
- Arm II (Waitlist Control [WLC]) (Active Comparator): Assessment including
  1. Wear an electronic accelerometer
  2. Quality of life assessment
  3. Physical fitness evaluation
  After waiting 6 months they will begin the fitness program as described in Arm I
  Interventions: Behavioral: Exercise Intervention; Behavioral: Internet-Based Intervention; Device: Monitoring Device; Other: Quality-of-Life Assessment

INTERVENTIONS:
Behavioral: Exercise Intervention — Participate in fitness program
Behavioral: Internet-Based Intervention — Engage in private social support messaging and Use the mobile app
Device: Monitoring Device — Wear an electronic accelerometer
  Other Names: Monitor
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This clinical trial studies a mobile health fitness program for adolescent and young adult childhood cancer survivors. Adolescent and young adult childhood cancer survivors are at risk to have negative late effects from treatment and to develop chronic health conditions. A sedentary lifestyle may increase the risk of cardiovascular disease, osteoporosis, and early mortality. Physical activity reduces the risk for cardiovascular disease and early mortality, improves cardiorespiratory fitness, muscular fitness, bone health, and body composition, and it is also positively associated with quality of life. Programs and technologies that promote physical activity are important because health behaviors adopted by adolescent and young adult childhood cancer survivors are likely to continue into adulthood. A mobile health fitness application may motivate adolescent and young adult childhood cancer survivors to engage and maintain physical activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of the technology-enhanced (electronic accelerometer + app + 8 weekly group sessions) fitness program in a pilot randomized clinical trial.

SECONDARY OBJECTIVES:

I. Determine the effectiveness of the technology-enhanced fitness program on participants' cardiorespiratory fitness and muscular fitness.

II. Examine the effects of the program on secondary outcomes of health related quality of life (HRQOL) and fatigue.

OUTLINE:

Participants are randomized to 1 of 2 arms.

ARM I (Intervention): Participants attend 8 group meetings weekly, wear an electronic accelerometer, engage in private social support messaging within the app and Facebook private groups, and then use the mobile app for 4 weeks without in-person groups.

ARM II (WAITLIST CONTROL [WLC]): After the 6 month assessment, participants receive the FitSurvivor intervention as in arm I.

ELIGIBILITY:
Inclusion Criteria:

* Any diagnosis of cancer prior to age 21
* Off treatment for at least 6 months
* For patients < 18 years, parents must give informed consent and patient must give assent; patients >= 18 must give informed consent

Exclusion Criteria:

* Any medical contraindication to exercise according to a physician or physician's designee
* Non-English speaking
* Current physical activity level exceeding Centers for Disease Control and Prevention (CDC) guidelines for activity (60 min of moderate-vigorous exercise/day for 5+ days/week (wk) including 3+ days of vigorous intensity activities and muscle-strengthening exercises on 3+ days/wk and bone strengthening exercises on 3+ days/wk for children < 18 and 150 min of moderate vigorous exercise or 75 min of vigorous exercise/wk and 2+ days of muscle strengthening activities for adults >= 18); the CDC guidelines are used to determine exercise prescription in our intervention; individuals already exceeding the guidelines would be unlikely to benefit from participating
* Significant developmental delay per patient, parent, or physician report
* Pregnant (per patient report); if participant becomes pregnant during the course of the study, she will be removed from further participation

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Devine, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 354 participants were mailed letters; 68 were contacted/screened, of which 56 were eligible and 49 enrolled (88% of those screened eligible, 14% of total potentially eligible pool).
Groups:
- Arm I (Intervention): Assessment including
  1. Wear an electronic accelerometer
  2. Quality of life assessment
  3. Physical fitness evaluation
  4. Participate in a fitness program which includes:
     * 8 group meetings over 90 minutes weekly
     * Behavioral internet based intervention engage in private social support messaging within the app and Facebook private groups and mobile app
  Exercise Intervention: Participate in fitness program
  Internet-Based Intervention: Engage in private social support messaging and Use the mobile app
  Monitoring Device: Wear an electronic accelerometer
  Quality-of-Life Assessment: Ancillary studies
- Arm II (Waitlist Control [WLC]): Assessment including
  1. Wear an electronic accelerometer
  2. Quality of life assessment
  3. Physical fitness evaluation
  After waiting 6 months they will begin the fitness program as described in Arm I
  Exercise Intervention: Participate in fitness program
  Internet-Based Intervention: Engage in private social support messaging and Use the mobile app
  Monitoring Device: Wear an electronic accelerometer
  Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Started | 25 | 24
Completed | 13 | 19
Not Completed | 12 | 5
Not completed — Lost to Follow-up | 11 | 5
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants in Group Qualitative, Group RCT ARM I and Group RCT Arm II, who completed any study activities after signing the consent form, are included. We excluded 2 participants (from Group Qualitative) who signed the consent form, but never completed qualitative interview.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC]) | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 12 | 25
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 18.88 [13 to 25] | 18.25 [13 to 25] | 18.56 [13 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 17 | 15 | 32
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Technology-enhanced Fitness Program
Description: Feasibility will be evaluated by the number of participants who enroll and complete baseline assessment for the randomized trial. In total, 354 participants were mailed letters; 68 were contacted/screened, of which 56 were eligible and 49 enrolled (88% of those screened eligible, 14% of total potentially eligible pool).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Intervention): Assessment including
  1. Wear an electronic accelerometer
  2. Quality of life assessment
  3. Physical fitness evaluation
  4. Participate in a fitness program which includes:
     * 8 group meetings of 90 minutes weekly
     * Behavioral internet based intervention engage in private social support messaging within the app and Facebook private groups and mobile app
  Exercise Intervention: Participate in fitness program
  Internet-Based Intervention: Engage in private social support messaging and Use the mobile app
  Monitoring Device: Wear an electronic accelerometer
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Number analyzed (Participants) | 25 | 24
Participants | 25 | 24

2. Secondary Outcome: Feasibility - Retention
Description: Percentage of participants who compete the 3 month assessment
Time Frame: Baseline to post-intervention (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Number analyzed (Participants) | 25 | 24
Participants | 15 | 22

3. Secondary Outcome: Fatigue Measured Using the PedsQL Multidimensional Fatigue Scale
Description: Fatigue measured using the PedsQL Multidimensional Fatigue Scale. The PedsQL Multidimensional Fatigue Scale yields three subscales: general, sleep/rest, and cognitive fatigue. Scores are transformed on a 0-100 scale, with higher scores indicating better functioning.
Time Frame: Baseline to post-intervention (3 months)
Population: Only participants with complete data were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Number analyzed (Participants) | 15 | 21
score on a scale
  Fatigue general (baseline) | 60.12 (25.72) | 71.02 (12.76)
  Fatigue general (post-intervention) | 65.18 (23.60) | 71.40 (13.44)
  Fatigue Sleep/Rest (baseline) | 55.95 (20.78) | 62.88 (15.90)
  Fatigue Sleep/Rest (post-intervention)) | 63.10 (24.78) | 65.72 (17.95)
  Fatigue Cognitive (baseline) | 57.74 (24.78) | 70.08 (22.59)
  Fatigue Cognitive (post-intervention) | 63.69 (26.27) | 75.38 (20.45)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effects of the intervention on changes in the General Subscale from baseline to post-intervention (3 months) were evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = 0.39, ANOVA; df = 33
Statistical Analysis 2: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effects of the intervention on changes in the Sleep/Rest Subscale from baseline to post-intervention (3 months) were evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = .49, ANOVA; df = 33
Statistical Analysis 3: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effect of the intervention on changes in the Cognitive Subscale from baseline to post-intervention (3 months) were evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = .83, ANOVA; df = 33

4. Secondary Outcome: Health Related Quality of Life (HRQL) Measured Using the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale
Description: The PedsQL Generic Core Scale is a well-validated measure of HRQOL with physical, emotional, social, and cognitive functioning domains. The PedsQL Generic Core yields two summary scores - Physical Summary and Psychosocial Summary. Scores are transformed on a 0-100 scale, with higher scores indicating better functioning.
Time Frame: Baseline to post-intervention (3 months)
Population: Only participants with complete data were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Number analyzed (Participants) | 15 | 21
score on a scale
  HRQOL: Physical Summary (baseline) | 72.10 (21.10) | 79.75 (8.32)
  HRQOL: Physical Summary (post-intervention) | 74.11 (20.74) | 81.68 (9.56)
  HRQOL: Psycho social Summary (baseline) | 72.64 (12.28) | 77.92 (12.14)
  HRQOL: Psycho social Summary (post-intervention) | 70.00 (16.17) | 75.92 (11.98)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effects of the intervention on changes in the PedsQL Physical Summary score were evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = .98, ANOVA; df = 33
Statistical Analysis 2: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effects of the intervention on changes in the PedsQL Psychosocial Summary score were evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = .85, ANOVA; df = 29

5. Secondary Outcome: Change in Cardiorespiratory Fitness Measured Using Submaximal Treadmill Test
Description: Cardiorespiratory fitness was measured via submaximal treadmill testing using a modified Bruce protocol. This standardized graded treadmill test adds two warm-up stages, with the first performed at a 1.7 mph and 0% grade and the second at 1.7 mph and 5% grade. Participants performed the graded exercise test until they reached 85% of their age-predicted maximum heart rate, which was measured using a chest-worn Polar heart rate monitor. Estimated VO2 max was calculated for each participant using the multi-stage model and American College of Sports Medicine metabolic equations.
Time Frame: Baseline to post-intervention (3 months)
Population: Only participants with complete data were included in this analysis.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Number analyzed (Participants) | 15 | 21
ml/kg/min
  estimated VO2 max (baseline) | 36.67 (7.03) | 40.61 (9.60)
  estimated VO2 max (post-intervention) | 39.08 (9.48) | 39.80 (9.27)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Test type: Superiority; p = .29, ANOVA; df = 29

6. Secondary Outcome: Change in Muscle Strength/Endurance Measured Using 10-repetition Maximum Strength Tests (Upper and Lower Body)
Description: Lower and upper body muscular strength/endurance were measured via 10-repetition maximum (10-RM) tests following National Strength and Conditioning Association guidelines (leg press machine for lower body and barbell bench press for upper body). Weight was increased until participants executed 10 repetitions in good form for both exercises. Estimates of 1-RM leg and bench press were made using a linear prediction equation. Higher scores indicate greater muscular strength/endurance.
Time Frame: Baseline to post-intervention (3 months)
Population: Only participant with complete data were included.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm I (Intervention) | Arm II (Waitlist Control [WLC])
Number analyzed (Participants) | 15 | 21
kg
  Lower Body 1-RM (baseline) | 191.93 (80.76) | 199.78 (84.56)
  Lower Body 1-RM (post-intervention) | 247.23 (109.76) | 219.71 (89.85)
  Upper Body 1-RM (baseline) | 35.78 (22.76) | 45.51 (25.83)
  Upper Body 1-RM (post-intervention) | 40.50 (24.26) | 48.48 (25.40)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effect of the intervention on changes in lower body estimated 1-RM was evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = .019, ANOVA; df = 32
Statistical Analysis 2: Comparison: Arm I (Intervention) vs Arm II (Waitlist Control [WLC]); Effect of the intervention on changes in upper body estimated 1-RM was evaluated using group x time in a repeated measures analysis of variance performed in SAS using PROC GLM for participants with complete data; Test type: Superiority; p = .34, ANOVA; df = 32

7. Secondary Outcome: Feasibility - Engagement With the App
Description: Engagement with the app was measured by 1) number of in-app exercises completed; 2) points earned (more active = more points); 3) achievements unlocked; and 4) number of likes and comments posted within the social feed. These are count data. Achievements unlocked has possible range of 0 to 20. Number of in-app exercises completed, points earned, and number of likes and comments posted within the social feed have a possible lower limit of 0 and no upper limit; higher numbers indicate more instances of each. The full range of participant data are: number of in-app exercises completed = 0-44; points earned = 0-1,195; number of achievements unlocked = 1-20; number of likes/comments posted = 0-8.
Time Frame: Duration of the FitSurvivor intervention (12 weeks)
Population: All participants from Arm I and Arm II who started the intervention were included. Those who dropped out prior to starting any sessions (n=7) were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: counts
Groups:
- ALL: Arm I (Intervention) and Arm II (WLC): All participants from Arm I and Arm II who started the 12-week intervention.
Arm/Group | ALL: Arm I (Intervention) and Arm II (WLC)
Number analyzed (Participants) | 42
counts
  # In-app workouts | 6.50 (10.69)
  Total in-app points earned | 165.48 (287.74)
  # Achievements unlocked | 8.50 (4.63)
  # of Likes/Comments posted | 0.62 (1.51)

ADVERSE EVENTS:
Time Frame: From the time first participant signed consent form until completion of all study related procedures. 3 years, 8 months.
Description: Project Coordinator maintains the adverse event log. All unexpected and/or serious adverse events occurring during the active portion of the intervention or up to 30 days after the last fitness program session, are reported to the Rutgers Cancer Institute of New Jersey Human Research Services and the Institutional Review Board. Adverse even log is also presented to Data Safety Monitoring Board for review.
Groups:
- Arm I (FitSurvivor Intervention): Assessment including
  1. Wear an electronic accelerometer
  2. Quality of life assessment
  3. Physical fitness evaluation
  4. Participate in a fitness program which includes:
     * 8 group meetings of 90 minutes weekly
     * Behavioral internet based intervention engage in private social support messaging within the app and Facebook private groups and mobile app
  Exercise Intervention: Participate in fitness program
  Internet-Based Intervention: Engage in private social support messaging and Use the mobile app
  Monitoring Device: Wear an electronic accelerometer
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm I (FitSurvivor Intervention) | Arm II (Waitlist Control [WLC])
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT02688192/Prot_SAP_000.pdf